CLINICAL TRIAL: NCT00863967
Title: Prospective Observational Cohort Study for Early Detection of Arteriosclerosis
Brief Title: Early Detection of Arteriosclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Barbara Biedermann MD, Department of medicine, Kantonsspital Bruderholz, CH-4101 Bruderholz
Other Study IDs: KSBH: 216/03
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Arteriosclerosis; Atherosclerosis; Myocardial Infarction; Stroke; Diabetes Mellitus; Peripheral Arterial Occlusive Disease
Keywords: physical examination; diagnostic techniques and procedures; diagnosis; immunologic tests; diagnostic tests; causality; genetic test; biomarker
MeSH Terms: conditions — Arteriosclerosis; Atherosclerosis; Myocardial Infarction; Stroke; Diabetes Mellitus; Peripheral Arterial Occlusive Disease 1; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood / serum / white cells / plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: no cardiovascular events
- 2: proven cardiovascular events
- 3: possible cardiovascular events

SUMMARY:
Arteriosclerosis is a common chronic disease with well known risk factors like diabetes mellitus, hypertension, dyslipidemia, adipositas and smoking, leading to severe complications like myocardial infarction, stroke or peripheral arterial occlusive disease. In addition to life-style factors there is also a genetic predisposition to develop complicated atherosclerosis.

Objective: Improve individual risk prediction by clinical phenotyping and genotyping.

DETAILED DESCRIPTION:
About 300 patients who are treated for various conditions at the department of general medicine at our hospital will be included prospectively in the study. This observational cohort will be followed for at least 10 years follow-up examinations.

At baseline and during follow up visits detailed clinical phenotyping is planned (medical and family history,standardized clinical and physical examinations, lab, RX, ECG, stress-test or echocardiogram). The genotyping is performed by DNA-isolation from leucocytes collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* informed consent

Exclusion Criteria:

* life-threatening disease
* life expectancy < 1 month
* uncapable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: teaching hospital primary care clinic
Sampling Method: Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2003-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 10 years at least

SECONDARY OUTCOMES:
Disease activity score | 2 / 5 / 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Biedermann, MD, Principal Investigator — Medical Department Kantonsspital Bruderholz CH-4101 Bruderholz

REFERENCES:
- [Background] Biedermann BC, Sahner S, Gregor M, Tsakiris DA, Jeanneret C, Pober JS, Gratwohl A. Endothelial injury mediated by cytotoxic T lymphocytes and loss of microvessels in chronic graft versus host disease. Lancet. 2002 Jun 15;359(9323):2078-83. doi: 10.1016/S0140-6736(02)08907-9. PMID 12086762
- [Background] Binder CJ, Chang MK, Shaw PX, Miller YI, Hartvigsen K, Dewan A, Witztum JL. Innate and acquired immunity in atherogenesis. Nat Med. 2002 Nov;8(11):1218-26. doi: 10.1038/nm1102-1218. No abstract available. PMID 12411948
- [Background] Kiechl S, Lorenz E, Reindl M, Wiedermann CJ, Oberhollenzer F, Bonora E, Willeit J, Schwartz DA. Toll-like receptor 4 polymorphisms and atherogenesis. N Engl J Med. 2002 Jul 18;347(3):185-92. doi: 10.1056/NEJMoa012673. PMID 12124407
- [Background] Nabel EG. Cardiovascular disease. N Engl J Med. 2003 Jul 3;349(1):60-72. doi: 10.1056/NEJMra035098. No abstract available. PMID 12840094
- [Background] Nakajima T, Schulte S, Warrington KJ, Kopecky SL, Frye RL, Goronzy JJ, Weyand CM. T-cell-mediated lysis of endothelial cells in acute coronary syndromes. Circulation. 2002 Feb 5;105(5):570-5. doi: 10.1161/hc0502.103348. PMID 11827921
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Stemme S, Faber B, Holm J, Wiklund O, Witztum JL, Hansson GK. T lymphocytes from human atherosclerotic plaques recognize oxidized low density lipoprotein. Proc Natl Acad Sci U S A. 1995 Apr 25;92(9):3893-7. doi: 10.1073/pnas.92.9.3893. PMID 7732003
- [Background] Strong JP, Malcom GT, McMahan CA, Tracy RE, Newman WP 3rd, Herderick EE, Cornhill JF. Prevalence and extent of atherosclerosis in adolescents and young adults: implications for prevention from the Pathobiological Determinants of Atherosclerosis in Youth Study. JAMA. 1999 Feb 24;281(8):727-35. doi: 10.1001/jama.281.8.727. PMID 10052443
- [Background] Yamada Y, Izawa H, Ichihara S, Takatsu F, Ishihara H, Hirayama H, Sone T, Tanaka M, Yokota M. Prediction of the risk of myocardial infarction from polymorphisms in candidate genes. N Engl J Med. 2002 Dec 12;347(24):1916-23. doi: 10.1056/NEJMoa021445. PMID 12477941